CLINICAL TRIAL: NCT02157272
Title: A Prospective, Randomized Clinical Trial Comparing Rivaroxaban vs Warfarin in High Risk Patients With Antiphospholipid Syndrome
Brief Title: Rivaroxaban in Thrombotic Antiphospholipid Syndrome
Acronym: TRAPS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unbalance in the composite endpoint between arms.
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Vittorio Pengo, Associate Professor of Cardiology, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2013-004575-13
Record Dates: First submitted 2014-05-31; First posted 2014-06-05 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Antiphospholipid Syndrome
Keywords: Antiphospholipid; Syndrome; Rivaroxaban; Warfarin; Thrombosis; Treatment
MeSH Terms: conditions — Antiphospholipid Syndrome; Syndrome; Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban 20mg qd, Rivaroxaban 15mg qd if creatinine clearance between 30-49 ml/min (calculated by Cockroft-Gault equation)
  Interventions: Drug: Experimental: Rivaroxaban
- Warfarin (Active Comparator): To Keep an INR between 2.0 and 3.0
  Interventions: Drug: Experimental: Rivaroxaban

INTERVENTIONS:
Drug: Experimental: Rivaroxaban — The investigated drug is Rivaroxaban 20mg, a film coated tablet, which is a highly selective direct factor Xa inhibitor. It should be administered orally, every day at any time (always the same), with food. The treatment should be performed for all the treatment period.
  Other Names: Xarelto

SUMMARY:
Primary Study Objective(s) The primary objective is to demonstrate the non-inferiority of Rivaroxaban 20 mg (or 15mgqd in case of moderate renal insufficiency) versus warfarin (INR 2.0-3.0) with respect to the occurrence of the cumulative end point of incident acute thrombosis (arterial or venous) confirmed by appropriate imaging studies, major bleedings, and death in triple aPL-positive APS patients.

Study Design A multicentre, interventional, prospective, parallel, randomised, controlled, open-label, Rivaroxaban 20 mg qd (or 15mg qd in patients with moderate renal insufficiency) vs warfarin (INR target 2.5), non-inferiority study, in 535 triple aPL-positive APS patients in approximately 40 Internal Medicine and Thrombosis centres. Each local Institutional Review Board will approve the study.

Study Population Patients of both sexes, of age 18-75, affected by anti-phospholipid syndrome, with a high probability of recurrences as defined by triple aPL-positivity, are eligible for this study.

Primary Outcome variables The primary cumulative outcome measure will be incident acute thrombosis (arterial or venous) confirmed by appropriate imaging studies, major bleeding, or death.

Secondary Outcome variables Separate evaluation of arterial and venous thrombosis and all-cause death.

04.27.2015: An amendment has been made. Enrollment permitted till 75 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form
2. Male or female of age 18-75 years
3. Triple aPL-positivity in the last blood sampling defined as:

   * aCL IgG/M (≥40 GPL or MPL, medium-to-high titer, and/or greater than the 99th percentile) and
   * aB2GPI IgG/M (≥40 U, medium-to-high titer, and/or greater than the 99th percentile) and
   * LA test positive based on the International Society of Thrombosis & Hemostasis Recommendations.
   * Positivity of aCL and abeta2GPI must be of the same isotype.
   * To confirm triple positivity for aPL and to validate the laboratory diagnosis, plasma (at least 2ml prepared by double centrifugation at 2000g) from patients of each Center will be stored at -80°C and later on sent in dry ice and retested in a reference laboratory (Padua Thrombosis Centre). Expenses for shipment will be in charge to the coordinator Center.
4. History of thrombosis (objectively proven arterial, venous, and/or biopsy proven microthrombosis) and/or pregnancy morbidity according to Miyaki

Exclusion Criteria:

Subjects meeting any of the following criteria will not be enrolled in the study:

1. Severe hypersensitivity reaction to rivaroxaban
2. Calculated CLCR <30 mL/min at the screening visit
3. Current pregnancy or breast feeding. Pregnancy is highly discouraged in these patients and if programmed patients are excluded from the study. If sexually active, be practicing an effective method of birth control (e.g., intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study
4. Concomitant treatment with other anticoagulants, such as unfractionated heparin, low molecular weight heparins (enoxaparin, dalteparin, etc.) heparin derivatives (fondaparinux), other oral anticoagulants (dabigatran etexilate, apixaban) in the case they can not be substituted with the study drugs.
5. Patients taking interfering medications: pharmacologic interactions may occur with strong inhibitors of p-glycoprotein and of CYP3A4, e.g., azole-antimycotics, such as ketoconazole, itraconazole, voriconazole, posaconazole, and HIV protease inhibitors; coadministration of rivaroxaban is therefore contraindicated in these cases. Several drugs used in neurological patients, such as phenobarbital, phenytoin, carbamazepine, and st john's wort (hypericum), are p-glycoprotein inducers and should be avoided. Whenever possible, it would be better to use levetiracetam and topiramate as antiepileptic therapy.
6. Hemorrhage Risk-Related Criteria

   * History of or condition associated with increased bleeding risk including, but not limited to:
   * Major surgical procedure or trauma within 30 days before the randomization visit
   * Clinically significant gastrointestinal bleeding within 6 months before the randomization visit
   * History of intracranial, intraocular, spinal, or atraumatic intra-articular bleeding
   * Chronic hemorrhagic disorder
   * Known intracranial neoplasm, arteriovenous malformation, or aneurysm
   * Planned invasive procedure with potential for uncontrolled bleeding.
   * Sustained uncontrolled hypertension: systolic blood pressure ≥180 mmHg
7. Known liver cirrhosis or ALT above three times the upper normal value.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-12; Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Cumulative outcome measure will be incident acute thrombosis (arterial or venous) confirmed by appropriate imaging studies, major bleeding, or death. | up to 4 years

SECONDARY OUTCOMES:
• Any single type of thromboembolic event | up to 4 years
All-cause mortality | up to 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Padua, Italy

REFERENCES:
- [Derived] Pontara E, Bison E, Cattini MG, Tonello M, Denas G, Pengo V. Close link between antiphosphatidylserine/prothrombin antibodies, lupus anticoagulant, and activated protein C resistance in tetra antiphospholipid antibody-positive subjects. J Thromb Haemost. 2023 Nov;21(11):3138-3144. doi: 10.1016/j.jtha.2023.06.033. Epub 2023 Jul 7. PMID 37422199
- [Derived] Pengo V, Denas G, Zoppellaro G, Jose SP, Hoxha A, Ruffatti A, Andreoli L, Tincani A, Cenci C, Prisco D, Fierro T, Gresele P, Cafolla A, De Micheli V, Ghirarduzzi A, Tosetto A, Falanga A, Martinelli I, Testa S, Barcellona D, Gerosa M, Banzato A. Rivaroxaban vs warfarin in high-risk patients with antiphospholipid syndrome. Blood. 2018 Sep 27;132(13):1365-1371. doi: 10.1182/blood-2018-04-848333. Epub 2018 Jul 12. PMID 30002145
- See also: Related info — http://www.dctv.unipd.it